CLINICAL TRIAL: NCT06760832
Title: How to Optimize Enteral Feeding of the Full Enteral Feeding Preterm Infant: Evaluation of Different Gastric Tube Management Practices
Brief Title: How to Optimize Enteral Feeding of the Full Enteral Feeding Preterm Infant
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: NE_PRE_20
Record Dates: First submitted 2024-12-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Preterm Birth; Feeding Methods
Keywords: enteral feeding; preterm newborns; full enteral feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Very low-birth-weight premature infants (VLBWs) are fed via nasal or oro-gastric tube for a long time because of the physiological inability to coordinate swallowing, sucking, and breathing until at least 34 weeks of gestational age.

Both bolus and continuous feeding modes are widely described in the literature; both modes have specific risks and benefits, and there is no evidence in the literature as to which mode is best in terms of tolerance and adverse effects.

To date, the characteristics of enteral feeding that are associated with better feeding tolerance and fewer adverse effects have not been uniquely documented.

There are currently no data in the literature directly comparing different modes of enteral feeding tube management in the preterm VLBW infant. Therefore, our study aims to evaluate different modes of enteral feeding tube management (extemporaneous vs. permanent introduction/removal and oral vs. nasal introduction route) in order to optimize enteral feeding management of the VLBW infant.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the tolerance of intermittent gastric tube placement versus permanent gastric tube maintenance in preterm VLBW infants who have achieved full enteral feeding, and to record the incidence of adverse effects associated with the different modes of gastric tube management.

Specifically, during bolus feeding, the following parameters will be evaluated in association with the two different management modes:

1. Presence, extent and characteristics of episodes of gastric stagnation
2. Incidence of cardio-respiratory events (desaturation and/or bradycardia)
3. Signs and symptoms of pain/discomfort related to the tube insertion and removal procedure In addition, the above parameters will be examined during enteral feeding with an orally or nasally introduced tube.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age <32 weeks and/or neonatal weight <1500 g
* Achievement of full enteral feeding (150 ml/kg/day of milk)
* Exclusive feeding of human milk (breast and/or bank)
* Informed consent signed by parent or legal guardian

Exclusion Criteria:

* Need for invasive ventilatory support
* Congenital malformations affecting the gastrointestinal tract

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all preterm infants of gestational age <32 weeks and/or neonatal weight <1500 g born at sant'orsola hospital. Based on birth data of preterm infants with these characteristics, it is estimated that within one year, approximately 50 infants will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the tolerance to intermittent gastric tube placement versus permanent gastric tube maintenance in Very Low Birth Weight preterm infants who have achieved full enteral feeding | From the 1st patient enrolled, up to 50th patient enrolled
  tolerance of intermittent gastric tube placement versus permanent gastric tube maintenance in preterm VLBW infants

CONTACTS AND LOCATIONS:
Overall Officials: Arianna Aceti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bolgona, Italy